CLINICAL TRIAL: NCT01568268
Title: A Randomized, Double Blind, Multicenter Phase III Trial to Evaluate the Therapeutic Efficacy and Safety of Palonosetron in Treatment of Postoperative Nausea and Vomiting
Brief Title: Therapeutic Efficacy and Safety of Palonosetron in Treatment of Postoperative Nausea and Vomiting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-11-112; CJ_ALX_302 (Other: CJ Cheiljedang Corporation)
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Laparoscopic Gynecologic, Abdominal, Other Surgery; General Anesthesia
Keywords: palonosetron; postoperative nausea and vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Palonosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palonsetron (Experimental)
  Interventions: Drug: Palonosetron
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo control group

INTERVENTIONS:
Drug: Palonosetron — palonosetron 0.075 mg intravenous injection over 10 seconds when nausea with NRS >= 4, or developement of retching or vomiting more than one time within three hour after the end of surgery.
  Other Names: Aloxi (palonosetron)
  Arms: Palonsetron
Drug: placebo control group — placebo intravenous injection over 10 seconds when nausea with NRS >= 4, or developement of retching or vomiting more than one time within three hour after the end of surgery.
  Other Names: placebo
  Arms: Placebo

SUMMARY:
This study was designed to evaluate the treatment efficacy and safety of palonosetron for the patients who undergo laparoscopic gynecologic, abdominal or other surgery under general anesthesia.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is a frequent complication of surgery, which can produce subject discomfort with medical and economic consequences. This study was designed to evaluate the treatment efficacy and safety of palonosetron for the subjects who undergo gynecologic or simple laparoscopic surgery. As the previous studies of palonosetron evaluated only the prevention of postoperative nausea and vomiting (PONV), there was no evidence-based guideline of palonosetron for treatment of PONV. The aim of the present study is to evaluate the treatment efficacy and safety of palonosetron for the patients who undergo laparoscopic gynecologic, abdominal or other surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 19 years and older, younger than 70 years old
* American society of Anesthesiologists physical status classification I to III
* those who undergo laparoscopic gynecologic, abdominal or other surgery under general anesthesia
* surgery for which anesthesia is expected to last at least 30 minutes
* if a subject has or may develop prolongation of cardiac conduction intervals, particularly corrected QT interval, he/she may be enrolled at the discretion of the investigator.

Exclusion Criteria:

* known hypersensitivity/ contraindication to 5-hydroxytryptamine antagonists or study drug excipient
* inability to understand or cooperate with the study procedures as determined by the investigator
* women who are pregnant, nursing or planning to become pregnant, are not using effective birth control, or that have had a positive serum pregnancy test within 7 days prior to surgery day 1.
* has received any investigational drug within 30 days before study entry
* having taken any drug with potential antiemetic efficacy within 24 hour prior to anesthetic procedures.
* any vomiting, retching, or nausea in the 24 hours preceding the administration of anesthesia
* known or suspected current history of alcohol abuse or drug abuse.
* any condition, which in the opinion of the investigator would make the subject ineligible for participation in the study

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Complete response at 24 hr | at 24 hour after randomization
  Complete response means no retching or vomiting and no administration of secondary rescue drug.

SECONDARY OUTCOMES:
Complete response at 72 hr | at 72 hour after randomization
  Complete response means no retching or vomiting and no administration of secondary rescue drug.
Complete control at 72 hr | at 72 hour after randomization
  Complete control means no retching or vomiting and no nausea with numerical rating scale >= 4 and no administration of secondary rescue drug.
Complete control at 24 hr | at 24 hour after randomization
  Complete control means no retching or vomiting and no nausea with numerical rating scale >= 4 and no administration of secondary rescue drug.
the incidence of nausea, retching, vomiting | at 24, 48, 72 hr after randomization
  the incidence of nausea with numerical rating scale >= 4, retching, vomiting
Time to recovery of nausea, retching, or vomiting | at 24, 48, 72 hr after randomization
  Time to recovery of nausea, retching, or vomiting from administration of palonosetron
the severity of nausea | at the time of, 24, 48, 72 hour after randomization
  the severity of nausea measured by NRS (numerical rating scale)
the incidence of rescue drug use | at 24, 48, 72 hour after randomization
  the incidence of rescue drug use
QOL by modified Osoba Nausea and Emesis Module | at 24, 48, 72 hour after randomization
  QOL by modified Osoba Nausea and Emesis Module

CONTACTS AND LOCATIONS:
Overall Officials: Tae Soo Hahm, MD, PhD, Study Director — Samsung Seoul Hospital, Samsung Medical Center; Youn Hong Kim, MD, PhD, Principal Investigator — Kangpook Samsung Hospital, Samsung Medical Center; Jung Won Hwang, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital; Joun Heum Yeon, MD, PhD, Principal Investigator — Sange Bahk Hospital, Inje School of Medicine
Locations (4):
- South Korea (4):
  - Samsung Medical Center, Seoul, Seoul
  - Bungdang Seoul National University Hospital, Seoul
  - Kangpook Samsung Hospital, Seoul
  - Sangye Bahk Hospital, Inje School of Medicine, Seoul

REFERENCES:
- [Derived] Hahm TS, Hwang JW, Kim WH, Oh EJ, Kim DK, Choi WJ, Kim YH, Ryu JH, Yoo BH, Yon JH. A prospective, randomized, double-blind, multicenter trial to evaluate the therapeutic efficacy and safety of palonosetron in the treatment of postoperative nausea and vomiting over a 72-h period. J Anesth. 2015 Feb;29(1):21-8. doi: 10.1007/s00540-014-1884-9. Epub 2014 Jul 19. PMID 25037960